CLINICAL TRIAL: NCT00431561
Title: Multi-national, Open-label, Active-controlled, Randomized Dose-finding Study to Evaluate Efficacy of 2 Doses of AP 12009 in Recurrent Glioma, Administered Intratumorally as Continuous High-flow Microperfusion Over 7 Days Every Other Week
Brief Title: Phase IIb Clinical Trial With TGF-β2 Antisense Compound AP 12009 for Recurrent or Refractory High-grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isarna Therapeutics GmbH (Industry)
Responsible Party: Hubert Heinrichs, MD, PhD, Chief Medical Officer, Antisense Pharma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP 12009-G004
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Glioblastoma; Anaplastic Astrocytoma
Keywords: Glioblastoma; Anaplastic astrocytoma; Antisense; Cancer; Transforming growth factor beta2 (TGF-beta2); Targeted therapy; Immunotherapy; Brain tumor; Central nervous system (CNS); Convection-enhanced delivery (CED) / microperfusion; Locoregional application
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Neoplasms; Brain Neoplasms; Camurati-Engelmann Syndrome | interventions — Trabedersen; Temozolomide; Lomustine; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AP 12009 10 µM (Experimental)
  Interventions: Drug: AP 12009 10 µM; Device: Drug delivery system for administration of AP 12009; Procedure: Placement of Drug Delivery System
- AP 12009 80 µM (Experimental)
  Interventions: Drug: AP 12009 80 µM; Device: Drug delivery system for administration of AP 12009; Procedure: Placement of Drug Delivery System
- Chemotherapy (Active Comparator)
  Interventions: Drug: temozolomide or PCV

INTERVENTIONS:
Drug: AP 12009 10 µM — 10 µM AP 12009 (trabedersen), intratumoral infusion, every other week, 11 cycles, maximum 21 weeks
  Arms: AP 12009 10 µM
Drug: AP 12009 80 µM — 80 µM AP 12009 (trabedersen), intratumoral infusion, every other week, 11 cycles, maximum 21 weeks
  Arms: AP 12009 80 µM
Drug: temozolomide or PCV — temozolomide: capsules, up to 200 mg/sqm/day, 5 days per cycle; PCV (procarbazine, CCNU, vincristine): standard regimen
  Other Names: Temodar; Temodal; TMZ; lomustine; Cecenu; CeeNU
  Arms: Chemotherapy
Device: Drug delivery system for administration of AP 12009 — Drug delivery system for Convection Enhanced Delivery consists of a portable pump with drug reservoir and infusion line. Main implanted parts are the port access system and the intratumoral catheter.
  Arms: AP 12009 10 µM; AP 12009 80 µM
Procedure: Placement of Drug Delivery System — Surgery for placement of intratumoral catheter and subcutaneous port access system as per routine clinical practice. Stereotactical catheter placement controlled by CT.
  Arms: AP 12009 10 µM; AP 12009 80 µM

SUMMARY:
In this multinational dose finding Phase IIb study the efficacy and safety of two doses of AP 12009 compared to standard chemotherapy (temozolomide or PCV) is investigated in adult patients with confirmed recurrent high-grade glioma.

DETAILED DESCRIPTION:
The purpose of this study is to compare the safety and efficacy of two doses of AP 12009 and standard chemotherapy in adult patients with recurrent high-grade glioma (anaplastic astrocytoma [AA], WHO grade III; or glioblastoma [GBM], WHO grade IV). AP 12009 is a phosphorothioate antisense oligodeoxynucleotide specific for the mRNA of human transforming growth factor-beta2 (TGF-beta2). The growth factor TGF-beta plays a key role in malignant progression of various tumors by inducing proliferation, invasion, metastasis, angiogenesis and escape from immunosurveillance. It has been shown that in a number of tumor types the degree of TGF-beta production strongly correlates with tumor grade and stage. In patients with high-grade glioma, the TGF-beta2 overexpression is associated with disease stage, clinical prognosis and the immunodeficient state of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of recurrent or refractory high-grade glioma (anaplastic astrocytoma, WHO grade III; or glioblastoma, WHO grade IV)
* Supratentorial localization
* No more than two chemotherapy regimens including radiochemotherapy since primary diagnosis
* Eligible for either TMZ or PCV treatment
* Recovery from acute toxicity caused by any previous therapy
* Adequate organ functions
* KPS at least 70%

Exclusion Criteria:

* Tumor surgery within 2 weeks prior to study entry
* Radiation therapy within 8 weeks prior to study entry
* Chemotherapy within 4 weeks prior to study entry (nitrosureas: 6 weeks)
* No more than 3 mg/day dexamethasone (or equivalent) at baseline
* Prior TGF-beta targeted therapy or tumor vaccination
* Baseline MRI shows mass effect
* Known active infection with HIV, HBV, or HCV; acute viral, bacterial, or fungal infection
* Significant psychiatric disorders/legal incapacity or a limited legal capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2003-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate of two AP 12009 dose groups and control group assessed by the evaluation of tumor size on brain MRI scans

SECONDARY OUTCOMES:
Overall survival | overall
Overall survival | six- and twelve-month
Response rates | at 3, 8, 10, and 12 months (and during the prolonged follow-up period in six-monthly intervals, if applicable)
Progression-free survival | six-month
Time to progression
Time to response
Best of all response rates assessed by survival status and variation of tumor size on brain MRI
Change of quality of life and Karnofsky Performance Status (KPS) | at 3, 8, 10, and 12 months (and during the prolonged follow-up period in six-monthly intervals, if applicable)
Best of all response rates
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Bogdahn, MD, Principal Investigator — University of Regensburg, Dept. of Neurology, Germany
Locations (36):
- Austria (3):
  - Universitätsklinik Innsbruck; Abteilung für Neurochirurgie, Innsbruck
  - Landes-Nervenklinik Wagner-Jauregg, Linz
  - Kaiser Franz Josef Spital, Abteilung für Neurologie, Vienna
- Sarajishvili Institute of Clinical Neurology and Neurosurgery, Tbilisi, Georgia
- Germany (12):
  - Medizinische Klinik und Poliklinik mit Schwerpunkt Onkologie und Hämatologie, Charité Campus Mitte, Berlin
  - Klinik und Poliklinik für Neurologie, Cottbus
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Gießen, Neurochirurgische Universitätsklinik, Giessen
  - Universitätsklinikum Kiel, Klinik für Neurochirurgie, Kiel
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Neurochirurgie, Leipzig
  - Universitätsklinik Magdeburg, Klinik für Neurochirurgie, Magdeburg
  - Universitätskliniken Mainz, Neurochirurgische Klinik und Poliklinik, Mainz
  - Universitätsklinikum Münster, Klinik und Poliklinik für Neurochirurgie, Münster
  - Klinikum und Poliklinik für Neurologie, Universität Regensburg, Regensburg
  - Klinikum Saarbrücken, Neurochirurgie, Saarbrücken
  - Neurologische Universitätsklinik Tübingen, Tübingen
- India (8):
  - Department of Neurosurgery, Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Sree Chitra Tirunal Institute for Medical Sciences & Technology, Department of Neurosurgery, Trivandrum, Kerala
  - Manipal Hospital; Manipal Institute for Neurological Disorders, Bangalore
  - Department of Neurosurgery, National Institute of Mental Health and Neurosciences, Bangalore
  - Department of Medical Oncology, Nizam's Institute of Medical Sciences, Hyderabad
  - Department of Neurosurgery, LTMG Hospital & LTM Medical College, Mumbai
  - Department of Neurosurgery, Neurosciences Center, New Dehli
  - Department of Neurological Sciences, Christian Medical College & Hospital, Vellore
- Israel (3):
  - Soroka Medical Center, Neurosurgery Department, Beersheba
  - Rambam Medical Center, Neurosurgery Department, Haifa
  - Rabin Medical Center, Neurosurgery Department, Petah Tikva
- Russia (9):
  - Tcheliabinsk Regional Clinical Hospital; State Medical Institution for Prophylaxis and Treatment, Chelyabinsk
  - Republican Clinical Hospital of Ministry of Health of Tatarstan Republic, Kazan'
  - Burdenko Neurosurgery Research Institute, Moscow
  - Omsk State Medical Academy; State Educational Institution of Higher Professional Education, Omsk
  - Polenov Neurosurgery Research Institute, Saint Petersburg
  - Military Medical Academy named after I.S.M. Kirov, Neurosurgery Department, Saint Petersburg
  - Medical Center "XXI century", Saint Petersburg
  - State Institution of Healthcare, Samara Regional Clinical Hospital in the name of M.I. Kalinin, Samara
  - Sverdlovsk Regional Oncological Clinic, Yekaterinburg

REFERENCES:
- [Derived] Uckun FM, Qazi S, Hwang L, Trieu VN. Recurrent or Refractory High-Grade Gliomas Treated by Convection-Enhanced Delivery of a TGFbeta2-Targeting RNA Therapeutic: A Post-Hoc Analysis with Long-Term Follow-Up. Cancers (Basel). 2019 Nov 28;11(12):1892. doi: 10.3390/cancers11121892. PMID 31795071